CLINICAL TRIAL: NCT00000875
Title: Controlled Clinical Trial of Antiviral Cytotoxic T Lymphocyte (CTL) Infusion Following Combination Antiretroviral Drug Therapy for Asymptomatic HIV-1 Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Model: Parallel | Purpose: Treatment
Other Study IDs: SPIRAT 3
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2003-04

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Immunotherapy, Adoptive; T-Lymphocytes, Cytotoxic; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Diphenhydramine; Lymphocyte Count; Lamivudine; Zidovudine; Acetaminophen; aldesleukin

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Diphenhydramine hydrochloride
Drug: Lymphocytes, Activated
Drug: Lamivudine
Drug: Zidovudine
Drug: Acetaminophen
Drug: Aldesleukin

SUMMARY:
To evaluate the safety of anti-HIV CTL therapy in early stage patients and to verify the safety when combined with antiviral therapy with zidovudine/lamivudine/indinavir and low-dose interleukin-2 (IL-2). To compare the effects on plasma and cell-associated viral load following combination drug therapy with and without antiviral CTL in early-stage patients. To study in detail the immune effects of lowering viral burden with antiviral combination drugs with and without T cell infusion on antiviral CTL activity, viral suppression and proliferation, circulating T cell phenotype, T cell apoptosis, CD4 cell numbers, DTH reaction, and inflammatory cytokine levels.

In an HIV-infected person, there is an ongoing struggle between HIV replication and host immune control. In the past decade most therapeutic strategies have targeted the virus. This approach has been frustrated by viral mutation to evade drug sensitivity. Promising drugs have recently been approved and there are encouraging sustained results from combination antiviral chemotherapy. However, even the most potent drug regimens do not seem to be curative, may eventually lead to drug resistance and may not completely restore lost immune function. The addition of immune-based therapy to antiviral drugs may lead to better viral control.

DETAILED DESCRIPTION:
In an HIV-infected person, there is an ongoing struggle between HIV replication and host immune control. In the past decade most therapeutic strategies have targeted the virus. This approach has been frustrated by viral mutation to evade drug sensitivity. Promising drugs have recently been approved and there are encouraging sustained results from combination antiviral chemotherapy. However, even the most potent drug regimens do not seem to be curative, may eventually lead to drug resistance and may not completely restore lost immune function. The addition of immune-based therapy to antiviral drugs may lead to better viral control.

This study has 2 regimens of 8 patients each. Patients are randomized as to CTL infusion only. Patients are stratified by viral load (less than 10,000 copies/ml vs. greater than or equal to 10,000 copies/ml). All patients receive combination drug therapy with AZT/3TC/indinavir for 9 months at which time patients have the option of continuing their study regimen another year or changing therapy. Patients in the T cell treatment regimen (regimen 2) receive 2 infusions of ex vivo expanded autologous anti-HIV CTL at 3 and 6 months after beginning AZT/3TC/indinavir therapy. The second infusion is administered with low-dose sc IL-2 1 day before and 4 days following T cell infusion.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Serologically confirmed HIV-1 infection.
* CD4 count >= 400/mm3.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following conditions or symptoms are excluded:

* Symptoms of HIV-1 disease, except lymphadenopathy.
* Symptoms of cardiac disease.
* Evidence of clinical pulmonary disease.
* Significant medical disease.

Patients with any of the following prior conditions are excluded:

* History of symptoms of HIV-1 disease, except lymphadenopathy.
* Participation in another experimental AIDS treatment clinical trial within 4 weeks into entry.
* History of significant psychiatric disease.
* History of pancreatitis, history of neuropathy or neurotoxic drug therapy.
* History of serious allergies requiring either systemic steroid therapy or prior hospitalization.
* History of significant arrhythmia, infarction or heart failure. Immunomodulatory therapy such as steroids or cyclosporine, systemic chemotherapy or alpha-interferon.

Prior Medication: Exclusion:

* Past treatment with any protease inhibitor.
* History of neurotoxic drug therapy.

Risk Behavior: Excluded

* Patients with current substance abuse.
* Excessive alcohol intake.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ctr For Blood Research Inc, Boston, Massachusetts, United States